CLINICAL TRIAL: NCT02437630
Title: An Investigation Into the Pressure and Airflow/Volume Changes Which Accompany Partial Closure of the Larynx During Expiration in Patients With COPD and the Effect of Applying a Positive End Expired Pressure by Facemask on These Parameters
Brief Title: Intrinsic PEEP and Laryngeal Aperture in COPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RO2014LF017B
Record Dates: First submitted 2015-01-27; First posted 2015-05-07 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with COPD: Patients with COPD aged >40 years with Gold stage II as measured by standard lung function testing or worse and at least 10 pack year history of smoking who will have insertion of an oesophageal balloon to measure intra-thoracic pressure, fibre-optic laryngoscopy to observe movement of the larynx during respiration and facemask pneumotachograph measurement of airflow and volumes at the mouth. The facemask which will be used to deliver a positive airway pressure (continuous positive airways pressure(CPAP) This will provide face mask CPAP with variation of mouth pressure with CPAP
  Interventions: Procedure: Oesophageal balloon to measure intra-thoracic pressure; Procedure: Fibre-optic laryngoscopy; Other: standard lung function tests; Procedure: face mask CPAP; Procedure: variation of mouth pressure with CPAP; Other: facemask pneumotachograph
- normal subjects without copd: Subjects without COPD and normal lung function as measured by standard lung function tests who will have insertion of an oesophageal balloon to measure intra-thoracic pressure, fibre-optic laryngoscopy to observe movement of the larynx during respiration and facemask pneumotachograph measurement of airflows and volumes at the mouth which will be used to deliver a positive airway pressure (continuous positive airways pressure CPAP) This will provide face mask CPAP with variation of mouth pressure with CPAP
  Interventions: Procedure: Oesophageal balloon to measure intra-thoracic pressure; Procedure: Fibre-optic laryngoscopy; Other: standard lung function tests; Procedure: face mask CPAP; Procedure: variation of mouth pressure with CPAP; Other: facemask pneumotachograph

INTERVENTIONS:
Procedure: Oesophageal balloon to measure intra-thoracic pressure — An oesophageal balloon will be inserted via a nostril after instillation of local anaesthetic and swallowed until the tip is in the lower third of the oesophagus. This will allow the intrathoracic pressure to be monitored via a pressure sensor attached to the oesophageal balloon catheter and placed next to the subject. This will allow us to observe the changes in oesophageal pressure during quiet breathing under a variety of applied positive pressure conditions.
Procedure: Fibre-optic laryngoscopy — A fibre-optic laryngoscope will be inserted through the opposite nostril to that used for the oesophageal balloon and placed with its tip abve the larynx where the laryngeal movement can be observed This will allow us to observe the changes in laryngeal aperture under a variety of applied positive pressure conditions.
Other: standard lung function tests — These will be carried out in any subject who has not had lung function testing in the previous 6 weeks and will be carried out by a lung function physiologist from the institution in accordance with standard procedures for lung function testing
Procedure: face mask CPAP — The subjects will wear a facemask with apertures for the oesophageal balloon and fibre-optic devices to cover the mouth and nose. airflow and volume will be recorded with a pneumotachograph and there will be tubing to connect to a positive pressure source (CPAP) to allow mouth pressures to be altered between 0-15cm H20.( 1cm H20 is the pressure produced by a column of water of 1centimetre in depth)
Procedure: variation of mouth pressure with CPAP — Once the other procedures are completed the subject will have his mouth pressure varied via application of positive pressure via a commercial CPAP device as used for treatment of obstructive sleep apnoea. The pressure will be varied randomly between 0-15cm H2O (water)for periods of 5 minutes both sitting and lying. Oesophageal balloon recording of intra-thoracic pressure and laryngeal movement and mouth airflow and volume will be recorded simultaneously and at the end of each 5 minute period the subject will be requested to take as big a breath in as possible to allow measurement of functional residual capacity and inspiratory capacity. This will allow us to observe the effect of changing mouth pressure with CPAP on laryngeal aperture and oesophageal pressures and airflow.
Other: facemask pneumotachograph — The facemask will incorporate a pneumotachograph to allow measurement of airflow and volumes throughout the respiratory cycle. This will allow us to observe the pattern of airflow with varying applied CPAP

SUMMARY:
In this study the investigators aim to investigate the extent to which in patients with chronic obstructive pulmonary disease narrowing of the vocal cords causes a positive pressure within the airways thus improving airflow and lung function. This information will be captured in the upright and lying down positions and an estimate of the magnitude of the effect will be formed by offsetting the pressure by asking the patients to breathe using a commercially available device used to treat sleep apnoea called a CPAP machine. This is an observational study in which the observation of laryngeal aperture, and mouth and oesophageal pressure at differing levels of applied CPAP will be recorded for analysis in patients with COPD and in normal subjects without COPD. All will have the same measurements, observations, and interventions to allow us to observe and measure pressure, laryngeal aperture, and airflow .

DETAILED DESCRIPTION:
In patients with chronic obstructive pulmonary disease (COPD) flow limitation inherent to the condition causes gas trapping and consequently over-inflation of the lung termed hyperinflation which worsens on exercise. Expiratory airflow can be maximized if the intrinsic positive pressure in the lung (Positive end expired pressure,PEEP) is offset by externally applied pressure (Expiratory positive airway pressure,EPAP) and it has been noted that patients with COPD do this by pursed lips breathing on expiration. The applicants have shown in a preliminary study that patients with COPD also close their vocal cords during expiration and is hypothesised that the function of the glottic narrowing was to provide an external positive expiratory pressure thus reducing flow limitation.

Relatively few data exist on laryngeal airflow in humans. One therapy that is increasingly used in the treatment of acute and chronic respiratory failure is non invasive pressure ventilation. Devices used for this oscillate between a high Inspiratory positive airway pressure (IPAP) and a lower Expiratory positive airway pressure (EPAP) but there remains uncertainty as how best to titrate the EPAP. We speculate that the optimum EPAP would be one to most reduce glottic narrowing on the basis that this would optimise expiratory flow and reduce the drive to glottic narrowing. The aim of this study is to test this hypothesis and to identify the range of external applied EPAP which minimises glottic narrowing in COPD patients in the erect and supine positions.

Technical advances with the use of continuous laryngoscopic examination (CLE) now provide a feasible and safe method to directly observe laryngeal movement from a fixed position. We aim to measure intra-thoracic pressure using an oesophageal balloon during respiration and to relate this to the CLE movement of the larynx.

At the same time we will be measuring airflow and volume with a pneumotachograph. This will allow us to identify the effect of glottic narrowing on intra-thoracic pressure and to see if the glottic narrowing does lead to an increased positive end expired pressure in the chest ( positive end expired pressure intrathoracic,PEEPi) and the extent to which it can be offset using EPAP delivered by a positive pressure machine (continuous positive airways pressure,CPAP).

The design of this study is a one visit physiological study which is an observational study with no blinding of investigator or participants.

We intend to study 10 controls with normal lung function and no history of COPD and 20 patients with COPD. They will attend for a single 3 hour period which will start with full explanation of the procedures to be undertaken and informed consent will be obtained on all aspects of the investigation by one of the investigators who is fully trained to obtain consent in research projects.

The subjects will be examined and have lung function tests if they have not already been carried out in the previous 6 weeks

The subject will be seated in an armchair and after application of local anaesthetic to the nose will be assisted to swallow an oesophageal balloon catheter in a deflated state inserted via a nostril and assisted by sipping water whilst the balloon is swallowed. The position of the balloon will be identified by measuring the length swallowed and positioned to the lower third of the oesophagus. A small quantity of air will be introduced into the balloon (1.0ml) to inflate the balloon and the tubing connected to a pressure measuring device situated next to the chair.

Next the subject will have introduced into their other nostril a fibre-optic laryngoscope which will be passed under direct vision to the back of the throat where the larynx in movement can be seen The output from the laryngoscope will be recorded digitally.

The subject will place over their mouth and nose a modified facemask through which they will be able to breathe without difficulty modified to admit the measurement catheters above. Attached to the mask will be a pneumotachograph which measures airflow and tubing to allow the pressure at the mouth to be varied.

This will allow the movement of the larynx on quiet breathing at rest to be observed with intra-thoracic pressure measured at the same time and the airflow at the mouth recorded simultaneously.

Once the subject is comfortable with these devices and relaxed in the chair recording of the laryngeal movement , pressures and airflow will be commenced and continue for 5 minutes. At the end of this time the subject will be asked to make an inspiratory capacity manoeuvre (breathe in as far as they can).

Subsequently the mouth pressure will be varied by 1cm H2O(1cm H20 = pressure produced by a column of water of 1cm depth) increments in random order 0-15cm H2O with 5 minutes at each level.

The protocol will then be repeated with the subject lying flat after which the catheter and the laryngoscope will be withdrawn.

Data will be stored securely in accordance with the Royal Brompton Hospital information governance and security protocols and access to personal data will only be by members of the research team. We will seek permission from the participants to inform their general practitioner or any other health professionals.

All data will be handled in accordance with the United Kingdom(UK) data protection Act 1998 and the condition of the main Research Ethics Committee (REC) approval.

The UK National Health Service Indemnity Scheme will meet any potential liability of the sponsors to harm to participants arising from the management of the research. any adverse events will be recorded in the case notes and a case report form and any serious adverse events will be reported to the study sponsor and the research ethics committee.

ELIGIBILITY:
Inclusion Criteria:

* patients with COPD
* Gold stage 11 as severity of disease
* aged 40+
* male and female
* at least 1 pack/day of cigarettes for >10 years
* normal subjects
* no evidence of Chronic Obstructive pulmonary disease (COPD) on spirometry
* < 1 pack of cigarettes/day for 10 years
* age >40
* male and female

Exclusion Criteria:

* an inability to comprehend what is proposed or travel to appointments
* restrictive lung pathology as assessed by history and lung function testing
* active infection
* evidence of cardiac disease
* inability to tolerate any of the following
* the fibre-optic laryngoscope
* the passing and retention of the oesophageal balloon
* the wearing of a face mask
* the application of a low level of positive pressure to the face mask and mouth ( CPAP, EPAP)
* those who are receiving a trial drug as part of another study at the time of study
* pregnancy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 20 patients with chronic obstructive pulmonary disease (COPD) Gold stage 11 as severity of disease aged 40+ male and female at least 1 pack/day of cigarettes for >10 years
  10 normal subjects no evidence of Chronic obstructive pulmonary disease (COPD) on spirometry < 1 pack of cigarettes /day for 10 years age >40 male and female
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
We will measure glottic aperture and compare glottic aperture observed with different levels of applied EPAP (expiratory positive airway pressure)in the erect and supine positions | 2 years
  we will measure glottic aperture and compare glottic aperture observed with different levels of applied EPAP on glottic opening in the erect and supine positions

SECONDARY OUTCOMES:
We will measure glottic aperture and and functional lung volumes ( inspiratory capacity and functional residual capacity) in the erect and supine positions at different levels of EPAP. | 2 years
  We will measure functional lung volumes , inspiratory capacity and functional residual capacity ,and the glottic aperture in the erect and supine positions at different levels of EPAP
We will determine the effect on PEEPi of applied EPAP in the erect and supine positions | 2 years
  We will determine the effect on PEEPi of applied EPAP in the erect and supine positions

CONTACTS AND LOCATIONS:
Overall Officials: michael Polkey, PhD, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- michael apps MD, London, United Kingdom